CLINICAL TRIAL: NCT02550340
Title: Munich Study for Beer Related ECG Change Workup
Acronym: Munich BREW
Status: Completed | Type: Observational
Sponsor: LMU Klinikum (Other)
Responsible Party: Principal Investigator, PD Dr. Stefan Brunner, Assistant Professor of Medicine, LMU Klinikum
Other Study IDs: Muc-M002-15
Record Dates: First submitted 2015-09-13; First posted 2015-09-15 (Estimated); Last update posted 2016-04-26 (Estimated); Status verified 2016-04

CONDITIONS: Arrhythmias, Cardiac
Keywords: Arrhythmia; Alcohol; ECG
MeSH Terms: conditions — Arrhythmias, Cardiac | interventions — Ethanol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Acute alcohol intake: Visitors of the Munich Octoberfest or similar events who fulfil in- and exclusion criteria
  Interventions: Other: acute alcohol intake

INTERVENTIONS:
Other: acute alcohol intake — Smart phone based ECG recording

SUMMARY:
The study aims to determine if acute recreational alcohol intake is associated with the occurence of ECG changes and arrhythmias.

DETAILED DESCRIPTION:
Both regular and acute excessive alcohol intake may deteriorate health. Possible sequelae include cardiac arrhythmias. For acute alcohol intake in particular it is insufficiently understood to what extent cardiac arrhythmias and other ECG changes occur, if the occurence depends on alcohol levels, and if there is a cut off value for occurence. Munich BREW aims to help clarifying these questions.

Participants of Munich BREW are identified and invited as visitors of the Munich Octoberfest and similar events. Participants need to be 18 years of age and over and need to declare theri will to participate. Following enrollment, participants will answer astudy questionnaire and will subsequently undergo recording of a 30 sec smart phone based ECG. Ultimately, the alcohol level is determined using a breath alcohol analyzer.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* informed conset signature

Exclusion Criteria:

* Incapability of contracting according to German law (BGB §105, paragraph 2)
* contraindications against ECG recording or alcohol breath test
* denial of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants of the Munich Octoberfest and similar events
Sampling Method: Non-Probability Sample
Enrollment: 3029 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Occurence of cardiac arrhythmias | 30 sec

SECONDARY OUTCOMES:
Alcohol related changes in ECG intervals | 30 sec

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Brunner, MD, Principal Investigator — LMU Klinikum
Locations (1):
- Klinikum der Universitaet Muenchen, Department of Medicine I, Munich, Germany

REFERENCES:
- [Derived] Brunner S, Drobesch C, Herbel R, Sinner MF. Effects of acute alcohol consumption on cardiac excitation, conduction, and repolarization: results from the Munich Beer Related Electrocardiogram Workup Study (MunichBREW). Clin Res Cardiol. 2021 Jun;110(6):916-918. doi: 10.1007/s00392-021-01839-6. Epub 2021 Mar 18. No abstract available. PMID 33738543
- [Derived] Brunner S, Herbel R, Drobesch C, Peters A, Massberg S, Kaab S, Sinner MF. Alcohol consumption, sinus tachycardia, and cardiac arrhythmias at the Munich Octoberfest: results from the Munich Beer Related Electrocardiogram Workup Study (MunichBREW). Eur Heart J. 2017 Jul 14;38(27):2100-2106. doi: 10.1093/eurheartj/ehx156. PMID 28449090